CLINICAL TRIAL: NCT05547230
Title: a Research About the Effect of Body Awareness on Work Motivation and Quality of Life, Among Primary School Teachers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Istanbul Arel University (Other)
Collaborators: sanem sener Assoc. Prof. PhD. (Unknown)
Responsible Party: Principal Investigator, Hasan Can Sogut, Research Assistant, Istanbul Arel University
Other Study IDs: 2022/13; İAÜ (Other: Istanbul Arel University)
Record Dates: First submitted 2022-03-23; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Quality of Life; Body Image; Motivation
Keywords: motivation; Quality of Life; Primary School; teachers
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- teachers: 4 basic components will be examined posture analysis body awareness work motivation quality of life
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — The same tests will be applied to all participants in an objective way.
  Other Names: posture analysis,body awareness,work motivation,quality of life questionnaires

SUMMARY:
The aim of this study is to investigate the effects of body awareness levels of teachers working in primary schools on work motivation and quality of life. In addition, the age, gender, height, weight, period of experience in the profession, smoking, branch, education level and current disease status of the teachers included in the study were also examined according to the questionnaire and evaluation scales. At the same time, the postures of the teachers were also evaluated.

The universe of the research consists of teachers working in public schools in Istanbul between April 2022 and September 2022. The sample, on the other hand, was determined as a total of 120 healthy volunteer teachers, 60 women and 60 men, who teach in 4 primary education institutions in avcılar and esenyurt districts of Istanbul.

Before starting the study, approval was obtained from the ethics committee of non-interventional clinical studies of Istanbul Arel University. Permission letters were obtained from the 4 primary education institutions where the study would be conducted and added to the ethics committee application form. The importance and purpose of the study were explained to all teachers who agreed to participate in the study. All necessary information was given on the subject that the results of the study would be used for scientific purposes, their identities would be kept confidential, and participants could withdraw from the study at any time, and their written consent was included in the informed consent form.

DETAILED DESCRIPTION:
This study is a descriptive cross-sectional study in which investigators will examine the effects of the body awareness levels of our teachers, who work in different institutions under different conditions, on their work motivation and quality of life, and also examine the posture of our teachers. After obtaining the necessary permissions from our volunteer teachers, the questionnaires and evaluation forms will be administered by a single therapist. Statistical analyzes will be made in SPSS, JASP, JAMOVI, R and Excel package programs, including sociodemographic data.

The body awareness of the teachers included in the study will be evaluated with the Body Awareness Questionnaire, their work motivation with the Job Motivation Scale, their quality of life with the Nottingham Health Profile questionnaire, and their posture assessment with the New York Posture Analysis method. In addition, the age, education level, experience, branch, body mass index, harmful habits and any diseases of the teachers participating in the study will be questioned and recorded. Questionnaires and measurements will be administered objectively by a single therapist.

A selection will be made from among the teachers who work in the educational institutions where permission is taken, who agree to be included in the study. All assessments will be performed by a single researcher during the study.

Face-to-face communication will be established with the participants by the responsible and assistant researcher in a way that will not affect the course hours.

According to the research, demographic data were obtained mainly with the Sociodemographic Information Form. its measurements were collected with body awareness, the Job Motivation Questionnaire, the Nottingham Health Profile Questionnaire, and the New York Posture, as evidenced by studies.

Participants, namely our teachers, will learn body awareness better with this study. At the same time, investigators think that participants will better understand the effects of body awareness levels on their working life and quality of life. Therefore, realizing that teachers, who are from the occupational group that has the most impact on the individual after the family, will have positive effects on students and society. The fact that the individuals who teach are good in every sense will lead to a better generation and a better society.

ELIGIBILITY:
Inclusion Criteria;

* be between the ages of 25-40
* Agree to participate in the study
* Approved for informed consent.
* Having worked actively for at least 1 year in the people who will participate in the study
* Having at least 6 months in the duty school to participate in the study

Exclusion Criteria;

* Being pregnant
* Presence of previous system migration
* Refusal to participate in the study
* 1 less assignment
* refusal to participate in the study

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Teachers between the ages of 25-40 working in Istanbul
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
To increase teachers' work motivation and quality of life by increasing their body awareness levels. | 3 months
  If teachers improve themselves, their success at school will also be high. The success of students will increase and it will be beneficial for social development.
  120 volunteer teachers aged 25-40 will be included in the study. Questionnaires and posture analysis will be made to teachers. all questionnaires will be administered at the beginning of the study . Statistical analyzes of the study will be made in SPSS, JASP, JAMOVI, R and Excel package programs.

CONTACTS AND LOCATIONS:
Overall Officials: sanem şener, 43, Principal Investigator — sanem.sener@beun.edu.tr
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Prof. Dr. Sebahattin Zaim Ilköğretim Okulu, Istanbul, Esenyurt
  - Istanbul Prof.Dr. Sebahattin Zaim Primary School, Istanbul, Esenyurt

IPD SHARING:
Plan to Share IPD: Undecided
After work the counselor will start with your teacher.

REFERENCES:
- [Background] Silva JPD, Fischer FM. Understudied school teachers' work/life balance and everyday life typologies. Chronobiol Int. 2020 Sep-Oct;37(9-10):1513-1515. doi: 10.1080/07420528.2020.1808010. Epub 2020 Aug 24. PMID 32835519
- [Background] Ellinger J, Mess F, Blaschke S, Mall C. Health-related quality of life, motivational regulation and Basic Psychological Need Satisfaction in Education Outside the Classroom: an explorative longitudinal pilot study. BMC Public Health. 2022 Jan 8;22(1):49. doi: 10.1186/s12889-021-12450-9. PMID 34998374
- See also: This study was conducted to investigate the relationship between body awareness, pain, emotional status, and quality of life among healthy people — https://www.journalagent.com/scie/pdfs/KEAH-20438-RESEARCH_ARTICLE-ALTUG.pdf